CLINICAL TRIAL: NCT06638996
Title: Psychological and Physiological Effects of Cannabigerol (CBG)
Brief Title: Acute Psychological and Physiological Effects of Cannabigerol
Acronym: CBG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington State University (Other)
Responsible Party: Principal Investigator, Carrie Cuttler, Associate Professor, Washington State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 20668-001
Record Dates: First submitted 2024-10-06; First posted 2024-10-15 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: No Disease or Condition is Being Studied
Keywords: CBG; Stress; Anxiety; Memory; Heart Rate; Electrodermal Activity; Cortisol; Blood Pressure; Pain
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The research assistants who administer the protocol will be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Arm (Placebo Comparator): Participants in this arm will receive a placebo
  Interventions: Other: Placebo Intervention
- CBG Arm (Experimental): Participants in this arm will receive CBG
  Interventions: Dietary Supplement: CBG Intervention

INTERVENTIONS:
Dietary Supplement: CBG Intervention — 50 mg CBG Administered
  Arms: CBG Arm
Other: Placebo Intervention — Participants will be administered a placebo
  Arms: Placebo Arm

SUMMARY:
The purpose of this study is to examine the acute effects of cannabigerol (CBG) on various psychological (e.g., anxiety, stress, mood, memory, impairment, intoxication, side effects) and physiological (blood pressure, cortisol, heart rate variability, electrodermal activity, pain tolerance, temperature) outcomes. Further, potential side effects of CBG (sleepiness/fatigue, dry mouth/eyes, increased appetite, and dizziness nausea) will be assessed. As such, the study is focused on better understanding some of the potentially beneficial and detrimental effects of CBG on humans.

DETAILED DESCRIPTION:
Recruitment: Healthy adult participants (aged 21+) will be recruited from the community via advertisements posted on campus, in businesses (including cannabis dispensaries), and on social media. Prospective participants will complete a brief online Qualtrics survey to determine eligibility. Specifically, to be eligible participants will need to be 21+ years of age, speak fluent English, be literate, be free of serious psychiatric disorders (psychotic disorders, bipolar disorders), neurological disorders (head injuries, brain tumors, Parkinson's disease), diabetes, low blood pressure, pregnancy, or breastfeeding. Participants must not report recent use (past 2 months) of illicit substances or dietary restrictions that would prevent them from eating the standardized breakfast (muffin, yogurt, juice/milk).

Eligible participants will be contacted via email and will be asked to schedule two testing sessions (1 week apart) that will begin between 8:00 and 9:30 am. They will be asked to abstain from CBG use for 1 week before the first testing session and to fast and abstain from cannabis use from midnight the night before each session (8 - 9.5 hours). The PI will use a random number generator to randomly assign each participant to ingest either the CBG tincture (50 mg) or placebo tincture orally in the first testing session and the opposite tincture in the second testing session.

Consent and Eligibility Confirmation. Participants will meet a graduate research assistant in The Health & Cognition (THC) lab in the Department of Psychology at Washington State University. After obtaining written informed consent participants will be asked when they last used CBG (if applicable), when they last used cannabis (if applicable), and when they last ate. Participants who report using CBG within the past week or cannabis after midnight the night prior or eating that day will be rescheduled and will be reminded that they must abstain from CBG for one week as well as from any cannabis use and food consumption on the day of the testing session. Participants who adhered to the abstinence requirements will be asked to complete a 12-panel urine drug test to ensure they test negative for illicit drugs. Participants who test positive for illicit drugs (other than THC) are not eligible and will not be permitted to complete the study. Participants who pass the drug test will have their blood pressure measured. Those with blood pressure lower than 90/60 mm Hg (indicating hypotension) will be excused.

T0 (Baseline) Assessments. Participants will be asked to wear a medical-grade wristband (Embrace device) that will continuously monitor their heart rate, electrodermal activity, and temperature. They will also be asked to provide a small saliva sample by rinsing their mouth for 1 minute, chewing on a Salivette for 1 minute, and then spitting the saturated Salivette in a sterile tube. Next, they will then complete a baseline assessment of motor/cognitive impairment using the DRiving Under the Influence of Drugs (DRUID) app.

Next, they will provide baseline ratings of their anxiety, stress, and mood using 0 to 10 visual analog rating scales. Participants will also rate their level of intoxication (to ensure it is 0) and provide baseline ratings of potential side effects (dry mouth, dry eyes, sleepiness, increased appetite, nausea, heart palpitations/racing heart, dizziness) using 0 (not at all severe) to 10 (extremely severe) visual analog scales. They will also be asked if they are experiencing any other physiological or psychological symptoms in an open-ended manner and to rate each on 0 (not at all) to 10 (severe) rating scales.

CBG/Placebo Administration. Once the baseline measures have been obtained, participants will be fed a high-fat (> 30g fat) breakfast (muffin, yogurt, milk/juice) to standardize food intake and increase the bioavailability/potency of the CBG. The research assistant will then give the participant the product (50 mg CBG or placebo) diluted in a small opaque cup of water to orally ingest in a double-blind manner (the PI will put the product in the testing room before each session). Next, participants will complete an online Qualtrics survey to measure demographic characteristics, depression, anxiety, and stress. They will then watch a 20-minute nature video to give the product additional time to take effect.

T1 Assessments. Approximately 25 minutes after product administration, participants will have their blood pressure measured, provide another saliva sample, and complete the DRUID impairment app. They will re-rate their anxiety, stress, and mood using 0 to 10 visual analog rating scales. They will also rate the drug effects (intoxication, drug effects, drug liking) and they will re-rate the potential side effects (dry mouth, dry eyes, sleepiness, increased appetite, nausea, heart palpitations/racing heart, dizziness). To capture other potential side effects, they will be asked if they are experiencing any other physiological or psychological symptoms in an open-ended manner and to rate the severity of each on 0 (not at all) to 10 (severe) rating scales.

T2 Assessments. Next, participants will engage in a modified version of the Maastricht Acute Stress Test (MAST) to determine whether CBG modifies responses to stress. Specifically, participants will complete three cold pressor trials in which they will be instructed to hold their hand in cold water (0 degrees) for 3 minutes. They will be informed they can remove their hand if it becomes too painful and the duration of time that they keep their hand in the cold pressor on each trial will be used as an objective measure of pain tolerance. After each trial, participants will subjectively rate the severity of pain they experienced using 0 to 10 visual analog rating scales. Between the three cold pressor trials, participants will be instructed to count backward from 2043 by 17s as quickly and as accurately as possible for 2 minutes. When they make an error, they will receive negative feedback and will be instructed to start the mental arithmetic over again. They will then rate their level of stress on a 0 (none) to 10 (extremely) scale.

After the MAST, participants will provide a third blood pressure assessment and saliva sample and will complete another trial of the DRUID app. They will re-rate their anxiety, stress, and mood using 0 to 10 visual analog rating scales. They will also re-rate subjective drug effects and side effects (using 0 to 10 visual analog rating scales and an open-ended question).

T3 Assessments. Next, participants will complete a short battery of memory tests. Specifically, they will complete the California Verbal Learning Test, the Deese-Roediger-McDermott paradigm, the Digit Span Forwards Test, and the Digit Span Backwards Test.

After the memory tests, participants will be asked to provide a fourth blood pressure assessment and saliva sample and will complete the DRUID app. They will re-rate their mood, anxiety, and stress. They will re-rate subjective drug effects and potential side effects including answering an open-ended question about perceived side effects with follow-up severity ratings.

Finally, participants will complete a brief survey to assess their cannabis and CBG use patterns.

Testing Session 2 After a one-week washout period participants will complete the second testing session which will be identical to the first session except for the product they will ingest. Specifically, those that ingested the 50 mg CBG tincture in Session 1 will ingest the 50 mg placebo tincture in Session 2 and those that ingested the placebo in Session 1 will ingest the CBG tincture in Session 2.

Alternate versions of the video, California Verbal Learning Test, and Deese-Roediger-McDermott paradigm will be administered in sessions 1 and 2 (in a counterbalanced manner).

ELIGIBILITY:
Inclusion Criteria:

21+ years of age Fluent in English

Exclusion Criteria:

Illiterate Serious psychiatric disorders (i.e., psychotic disorders, bipolar disorders) Intellectual disability Chronic neurological disorders (e.g., head injuries, brain tumors, Parkinson's disease) Diabetes Low blood pressure Pregnant or breastfeeding Recent illicit drug use (past 2 months) - does not include cannabis Dietary restrictions preventing them from eating muffin, yogurt, milk/juice

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-10-28 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Anxiety | Anxiety ratings will occur within a 2.5 hour time frame for each session with sessions scheduled approximately one week apart
  Anxiety will be assessed along a 0 to 10 rating scale at baseline (T0), ~40 minutes after ingesting placebo or CBG (T1), after the stress test (T2), and after the memory tests (T3). Change scores from baseline to each time point will be examined.
Stress | Stress ratings will occur within a 2.5 hour time frame for each session with sessions scheduled approximately one week apart
  Stress will be assessed along a 0 to 10 rating scale at baseline (T0), ~40 minutes after ingesting placebo or CBG (T1), after the stress test (T2), and after the memory tests (T3). Change scores from baseline to each time point will be examined.
Mood | Mood ratings will occur within a 2.5 hour time frame for each session with sessions scheduled approximately one week apart
  Mood will be assessed along a 0 to 10 rating scale at baseline (T0), ~40 minutes after ingesting placebo or CBG (T1), after the stress test (T2), and after the memory tests (T3). Change scores from baseline to each time point will be examined.
Salivary Cortisol | Saliva samples will be collected within the 2.5 hour time frame for each session with sessions scheduled approximately one week apart
  Salivary Cortisol will be collected using Salivettes at baseline (T0), ~40 minutes after ingesting placebo or CBG (T1), after the stress test (T2), and after memory the memory tests (T3). Change scores from baseline to each time point will be examined.
Electrodermal Activity | Electrodermal Activity will be measured continuously for the duration of the 2.5 hour session for each session with sessions scheduled approximately one week apart
  Electrodermal Activity will be assessed continuously using an Embrace wristband device from baseline to the end of the study. Primary points of interest include baseline (T0), after ingesting placebo or CBG (T1), after the stress test (T2), and after the memory tests (T3).
Heart Rate/Heart Rate Variability | Heart Rate/Heart Rate Variability will be assessed continuously for the duration of the 2.5 hour session with sessions scheduled approximately one week apart
  Heart rate/heart rate variability will be assessed continuously using an Embrace wristband device from baseline to the end of the study. Primary points of interest include baseline (T0), after ingesting placebo or CBG (T1), after the stress test (T2), and after the memory tests (T3).
Blood Pressure | Blood Pressure will be obtained multiple times throughout the 2.5 hour session for each session with sessions scheduled approximately one week apart
  Blood Pressure will be assessed at baseline (T0), ~40 minutes after ingesting placebo or CBG (T1), after the stress test (T2), and after the memory tests (T3). Change scores from baseline to each time point will be examined.
Pain Tolerance | Pain tolerance will be assessed within a 2.5 hour time frame for each session with sessions scheduled approximately one week apart
  Pain tolerance will be assessed by computing the duration of time they keep their hand in the cold pressor on each of the three cold pressor trials.
Verbal Memory | Participants will complete this test within a 2.5 hour time frame for each session with sessions scheduled approximately one week apart
  Participants will complete the California Verbal Learning Test
Short-Term/Working Memory | Participants will complete this test within a 2.5 hour time frame for each session with sessions scheduled approximately one week apart
  Participants will complete the Digit Span Forwards and Digit Span Backwards Tests
False Memory | Participants will complete this test within a 2.5 hour time frame for each session with sessions scheduled approximately one week apart
  Participants will complete the Deese-Roediger-McDermott paradigm.

SECONDARY OUTCOMES:
Impairment | Participants will complete the DRUID app within the 2.5 hour time frame for each session with sessions scheduled approximately one week apart
  Participants will complete the DRiving Under the Influence of Drugs (DRUID) app at baseline (T0), ~40 minutes after ingesting placebo or CBG (T1), after the stress test (T2), and after the memory tests (T3).
Subjective Drug Effects | Subjective drug effect ratings will occur within a 2.5 hour time frame for each session with sessions scheduled approximately one week apart
  Participants will provide ratings of their levels of intoxication, level of perceived drug effects, and drug liking using 0 -10 scales ~40 minutes after ingesting placebo or CBG (T1), after the stress test (T2), and after the memory tests (T3).
Side Effects | Side effect ratings will occur within a 2.5 hour time frame for each session with sessions scheduled approximately one week apart
  Participants will provide ratings of various side effects (dry eyes, dry mouth, increased appetite, racing heart/heart palpitations, nausea, dizziness) using 0-10 scales and they will be asked if they are experiencing any additional physiological or psychological symptoms in an open-ended manner and if applicable to rate these on 0 to 10 rating scales at baseline (T0), ~40 minutes after ingesting placebo or CBG (T1), after the stress test (T2), and after the memory tests (T3). Change scores from baseline to each time point will be examined.

CONTACTS AND LOCATIONS:
Locations (1):
- Washington State University - Pullman Campus, Pullman, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared upon request and after publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Deidentified data will be retained indefinitely
Access Criteria: Researchers wanting to conduct secondary data analysis following my own publication